CLINICAL TRIAL: NCT05549752
Title: Safety and Efficacy of Flecainide Versus Amiodarone in the Cardioversion of Paroxysmal Atrial Fibrillation at the Emergency Department, in Patients With Coronary Artery Disease Without Residual Ischemia and Ejection Fraction > 35%
Brief Title: Flecainide Versus Amiodarone in the Cardioversion of Paroxysmal Atrial Fibrillation at the Emergency Department, in Patients With Coronary Artery Disease Without Residual Ischemia
Acronym: FLECA-ED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Collaborators: Win Medica (Unknown); Pharmassist Ltd (Industry)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Principal Investigator. Prof. Konstantinos P. Tsioufis, MD, PhD, FESC, FACC, Professor of Cardiology, Director of 1st Department of Cardiology, Hippokratio Hospital, University of Athens, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLECA-ED
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation Paroxysmal; Coronary Artery Disease Without Residual Ischemia
Keywords: Flecainide; Amiodarone
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flecainide (Active Comparator)
  Interventions: Drug: Flecainide Injectable Solution
- Amiodarone (Active Comparator)
  Interventions: Drug: Amiodarone Injectable Solution

INTERVENTIONS:
Drug: Flecainide Injectable Solution — Intravenous Flecainide at a dose of 2.0mg/kg (maximum dose: 150mg) in 100ml D/W 5% for 10 minutes.
  Arms: Flecainide
Drug: Amiodarone Injectable Solution — Intravenous Amiodarone at a dose of 5.0-7.0 mg/kg for 1 hour, and maintenance dose of 50mg/h (maximum dose: 1000mg) for up to 24 hours.
  Arms: Amiodarone

SUMMARY:
Current guidelines for the cardioversion of paroxysmal Atrial Fibrillation at the Emergency Department do not prioritize between antiarrhythmic agents and do not consider the time taken for successful cardioversion. Furthermore, the use of flecainide -a class 1C antiarrhythmic agent- is contraindicated for the cardioversion of patients with revascularized coronary artery disease, as well as patients with ischemic cardiomyopathy and preserved ejection fraction. These recommendations stem from insufficient data, mainly from the CAST study.

The present study is a prospective, multicentre, randomized clinical trial. The primary goals of this clinical trial are to prove the superiority of flecainide over amiodarone in the successful cardioversion of paroxysmal atrial fibrillation at the Emergency Department, and to prove that the safety of flecainide is non-inferior to amiodarone, in patients with coronary artery disease without residual ischemia and ejection fraction over 35%. The secondary goals of the study are to prove the superiority of flecainide over amiodarone in the reduction of hospitalizations from the Emergency Department due to atrial fibrillation, in the time taken to achieve cardioversion, and to the reduction of the need to conduct electrical cardioversion.

The study population will be all consecutive new-comers to the Emergency Department with primary diagnosis of paroxysmal atrial fibrillation and history of coronary artery disease without angina, without residual ischemia and with ejection fraction > 35%. The sample size will be 200 patients, who will be monitored for 30 days. At the Emergency Department, all patients will be under continuous ECG monitoring, and a 24-hour ECG device will also be placed (Holter). The patients will be randomized to the treatment group (flecainide) and the control group (amiodarone).

Patients in both arms will stay at the ED for a total of 6 hours after therapy initiation. If no adverse events occur in this time, the patient will be discharged from the ED. Otherwise, the patient will be admitted to the hospital. At 24 hours, the patients will visit the study centre for physical examination, ECG, cardiac ultrasound, 24-hour ECG removal and adverse events evaluation. At 30 days, follow-up via phone calls will be conducted for the evaluation of the study outcomes and adverse events.

As of June 2025, an interim analysis has been completed, and preliminary study results have been submitted for presentation at the European Society of Cardiology (ESC) Congress. Based on the interim findings, the study's target sample size has been revised to a total of 80 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-85 years old
2. Paroxysmal Atrial Fibrillation, documented by 12-lead ECG, with one of the following:

   1. Atrial Fibrillation onset less than 48 hours from the time of presentation to the Emergency Department
   2. Atrial Fibrillation onset between 48 hours and 7 days from the time of presentation to the Emergency Department, and patient has been on anticoagulation for at least 30 days
   3. History of Coronary Artery Disease without residual ischemia, defined by one of the following criteria:

      * PCI <= 1 year, or
      * CABG <= 3 years, or
      * Negative imaging-based stress testing within 1 year, and:

        * History of known coronary artery stenosis > 60% without revascularization, or
        * PCI >= 1 year, or
        * CABG >= 3 years
3. Ejection Fraction > 35% (documented by cardiac ultrasound at the Emergency Department, or within 1 year)
4. Signed informed consent from the patient or legal representative.

Exclusion Criteria:

1. Based on ECG at the Emergency Department:

   1. Atrial Flutter
   2. Newly documented Left Bundle Branch Block (LBBB)
   3. Newly documented Right Bundle Branch Block (RBBB) with QRS duration > 150ms
2. Previously documented 24-hour ECG holter monitoring with > 720 poly PVCs/24hours, or non sustained ventricular tachycardia
3. No history of coronary artery disease
4. ST-Segment Elevation Myocardial Infarction (STEMI)
5. Non-ST-Segment Elevation Myocardial Infarction (NSTEMI), according to ESC 2020 guidelines on NSTEMI:

   1. If troponin at t0h is over the "low" criterion on table of the cutoff values
   2. If the change of troponin (Δtroponin) at t1h is over the respective cutoff value at the table for the cutoff values
6. Unstable angina, defined as myocardial ischemia at rest or at minimum effort, in the absence of acute injury/necrosis of myocardial cells
7. Known residual ischemia:

   1. Positive imaging-based stress testing
   2. Negative imaging-based stress testing >= 1 year, and:

      * History of known coronary artery stenosis > 60% without revascularization, or
      * PCI >= 1 year, or
      * CABG >= 3 years
8. History of acute coronary syndrome within 1 year
9. Severe Aortic Valve Stenosis (mean pressure gradient > 40mmHg, AVA < 1cm/m^2)
10. Severe Chronic Kidney Disease (stage >= 4)
11. Severe systematic disease, including neoplasmatic disease under any antineoplasmatic treatment, liver failure, infection with fever
12. Use of strategy "pill in the pocket", by taking flecainide (max 200mg) or propafenone (max 600mg) within 6 hours prior to Emergency Department visit
13. Known dysanexia or allergy to flecainide or amiodarone
14. Pregnancy or/and breastfeeding
15. Participation in any other clinical trial
16. Life expectancy less than 1 year
17. Inappropriate, unfit, or unwilling to follow the desingated protocol procedures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of successful cardioversion to sinus rhythm | From the drug initiation and for 6 hours
The combined frequency of premature ventricular contractions (PVCs), non-sustained ventricular tachycardia (NSVT), sustained ventricular tachycardia (SVT), bradycardia < 50bpm and systolic blood pressure < 90mmHg. | From the drug initiation and for 6 hours

SECONDARY OUTCOMES:
The frequency of patient discharges from the Emergency Department in sinus rhythm | From the drug initiation and for 6 hours
The frequency of successful cardioversion to sinus rhythm | From the drug initiation and for 24 hours, 24 hour ECG Holter monitoring
The time until the cardioversion to sinus rhythm | From the drug initiation and for 6 hours
The frequency of electrical cardioversion | From the drug initiation and for 24 hours
The frequency of arrhythmias: burden of PVCs, NSVT episodes, SVT episodes | From the drug initiation and for 24 hours
The frequency, severity and type of Adverse Events | From the drug initiation and for 30 days

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - First Department of Cardiology, Hippocration General Hospital, National and Kapodistrian University of Athens, Athens, Greece, Athens
  - Konstantopoulio General Hospital, Athens
  - KAT General Hospital, Athens

IPD SHARING:
Plan to Share IPD: No